CLINICAL TRIAL: NCT00978731
Title: Long-Term Safety and Efficacy of Dasatinib (BMS-354825) in Chronic Myelogenous Leukemia or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia in Subjects Who Experienced Clinical Benefit on Protocol CA180-002
Brief Title: Chronic Myelogenous Leukemia or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-039
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Dasatinib; src-Family Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, The dosing ranges from 50mg to a total of 240mg daily with the following 3 schedules:
  * 5 days on, 2 days off
  * 6 days on, 1 day off
  * Continuous daily dosing
  Once Daily (QD) or Twice Daily (BID) dosing, Subjects will be treated until progression of disease despite escalation/reductions of dose to the level deemed safe by available data, until intolerable/unacceptable toxicity or until subject withdrawal from the study or discontinuation of the study
  Other Names: BMS-354825; Sprycel; Src Kinase

SUMMARY:
To determine the long term safety and tolerability of dasatinib exposure in subjects previously treated in CA180-002.

ELIGIBILITY:
This study enrolled participants with Philadelphia chromosome positive (Ph+)chronic myelogenous leukemia (CML) or Ph+ acute lymphoblastic leukemia (ALL) who had demonstrated hematologic resistance or intolerance to imatinib mesylate (Gleevec) and had experienced clinical benefit (in Investigator's opinion) on protocol CA180002.

Inclusion Criteria:

* Signed written informed consent
* Previous treatment with dasatinib on protocol CA180-002 and receiving clinical benefit in the opinion of the investigator
* Completed a minimum of 3 months on protocol CA180-002
* Eastern Cooperative Oncology Group (ECOG)performance status 0, 1, or 2 (See Appendix 1)
* Prior history of Ph+ chronic, accelerated, or blast phase CML or Ph+ ALL

Exclusion Criteria:

* Women of childbearing potential(WOCBP)who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 12 weeks after the study
* WOCBP using a prohibited contraceptive method
* Women who are pregnant or breastfeeding
* Met the criteria as defined in protocol CA180-002 for discontinuation of therapy which includes:
* Withdrawal of informed consent (subject's decision to withdraw for any reason)
* Any clinical adverse event, laboratory abnormality or intercurrent illness which, in the opinion of the investigator, indicates that continued treatment with dasatinib is not in the best interest of the subject
* Imprisonment or the compulsory detention for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Medical History and Concurrent Diseases

* A serious uncontrolled medical disorder or active infection which would impair the ability of the patient to receive protocol therapy;
* Uncontrolled angina within 3 months
* Diagnosed or suspected congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Prolonged corrected QT(QTc) interval on pre-entry electrocardiogram (> 450 msec)
* Uncontrolled hypertension
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent;
* History of significant bleeding disorder unrelated to CML, including:

  1. Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  2. Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)

Physical and Laboratory Test Findings

* Total bilirubin ≥ 1.5 mg/dl
* alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 2 times the institutional upper limits of normal
* Serum creatinine ≥ 1.5 times the institutional upper limits of normal

Prohibited Therapies and/or Medications

* Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes including:

  * quinidine, procainamide, disopyramide
  * amiodarone, sotalol, ibutilide, dofetilide
  * erythromycins, clarithromycin
  * chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
* Medications that inhibit platelet function and any non-steroidal anti-inflammatory drug) or anticoagulants are prohibited unless a previous exception on CA180-002 was granted by the medical monitor. Subjects taking anagrelide for thrombocytosis due to CML are eligible for this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry: Participants with Chronic Myelogenous Leukemia (CML)were continued on the last dose and schedule of dasatinib that was received within the previous protocol CA180002 (NCT00064233). A total daily dose (TDD) of 50 mg, 75 mg, 105 mg, 140 mg or 180 mg dasatinib was taken once daily (QD). Participants were dosed on 1 of 3 schedules (5 days on, 2 days off; 6 days on, 1 day off or continuous daily dosing) and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
- CML: BID Dosing at Study Entry: Participants with CML were continued on the last dose and schedule of dasatinib that was received within the previous protocol CA180002 (NCT00064233). Treatment was received BID, with a TDD of 50 mg, 70 mg, 100 mg, 140 mg, 180 mg or 240 mg dasatinib. Participants were dosed on 1 of 3 schedules (5 days on, 2 days off; 6 days on, 1 day off or continuous daily dosing) and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
- Accelerated Phase CML: BID Dosing at Study Entry: Participants with accelerated phase CML were continued on the last dose and schedule of dasatinib that was received within the previous protocol CA180002 (NCT00064233). A TDD of 50 mg, 75 mg, 105 mg, 120 mg, 140 mg or 180 mg dasatinib was taken QD or split into 2 doses and taken BID (TDD of 50 mg, 70 mg, 100 mg, 140 mg, 180 mg or 240 mg). Participants were dosed on 1 of 3 schedules (5 days on, 2 days off; 6 days on, 1 day off or continuous daily dosing) and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
- Myeloid Blast Phase CML: BID Dosing at Study Entry: Participants with myeloid blast phase CML were continued on the last dose and schedule of dasatinib that was received within the previous protocol CA180002 (NCT00064233). A TDD of 50 mg, 75 mg, 105 mg, 120 mg, 140 mg or 180 mg dasatinib was taken QD or split into 2 doses and taken BID (TDD of 50 mg, 70 mg, 100 mg, 140 mg, 180 mg or 240 mg). Participants were dosed on 1 of 3 schedules: 5 days on, 2 days off; 6 days on, 1 day off; or continuous daily dosing and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
Period: Overall Study
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry
Started | 22 | 15 | 5 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 22 | 15 | 5 | 4
Not completed — Death | 4 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Adverse Event | 5 | 2 | 0 | 0
Not completed — Participant's request | 1 | 0 | 0 | 0
Not completed — Administrative reason | 3 | 3 | 1 | 0
Not completed — Deterioration without progression | 0 | 1 | 0 | 0
Not completed — Disease progression/relapse | 5 | 4 | 2 | 2
Not completed — Study closure | 3 | 4 | 1 | 1
Not completed — No response | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry | Total
Number analyzed (Participants) | 22 | 15 | 5 | 4 | 46
Age Continuous [Median (Full Range); unit: years] | 58 [41 to 81] | 68 [30 to 80] | 63 [51 to 74] | 51 [34 to 62] | 64 [30 to 81]
Age, Customized [Number; unit: participants]
  < 65 years | 12 | 5 | 3 | 4 | 24
  >= 65 years | 10 | 10 | 2 | 0 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 4 | 1 | 23
  Male | 11 | 8 | 1 | 3 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 18 | 11 | 3 | 3 | 35
  Black/African American | 2 | 3 | 1 | 0 | 6
  Asian | 0 | 1 | 0 | 0 | 1
  Other races | 2 | 0 | 1 | 1 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — The ECOG PS is used to assess disease severity, with 0 being the least severe score and 5 being the most severe score. A score of 0 is fully active; 1 is restricted physically strenuous activity; 2 is ambulatory but unable to work; 3 is capable of only limited self care; 4 is completely disabled; 5 is dead.
  participants
    0 = fully active | 18 | 13 | 3 | 4 | 38
    1 = restricted physically strenuous activity | 4 | 1 | 2 | 0 | 7
    2 = ambulatory but unable to work | 0 | 0 | 0 | 0 | 0
    3 = capable of only limited self care | 0 | 0 | 0 | 0 | 0
    4 = completely disabled | 0 | 0 | 0 | 0 | 0
    5 = dead | 0 | 0 | 0 | 0 | 0
    Not reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died, Experienced Other Serious Adverse Events (SAEs), Adverse Events (AEs) and AEs Leading to Study Drug Discontinuation.
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to AEs were recorded. These data differ from that in the Participant Flow section. This is because the data were collected on 2 different pages of the Case Report Form and were not reconciled.
Time Frame: From start of study until up to 30 days after end of study participation. Median duration of exposure (on-study time) was 23.4 months.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15 | 5 | 4
participants
  Deaths | 3 | 2 | 1 | 1
  SAEs | 10 | 9 | 3 | 3
  AEs | 22 | 15 | 5 | 4
  Discontinuation due to AEs | 4 | 3 | 1 | 0

2. Primary Outcome: Number of Participants Who Experienced Drug-related AEs and Drug-related SAEs.
Description: Drug-related AEs are those events with a relationship to the study therapy of certain; probable; or possible or missing. Drug-related SAEs are those events with any relationship to the study therapy.
Time Frame: as for outcome 1
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15 | 5 | 4
participants
  Drug-related AEs | 14 | 9 | 3 | 3
  Drug-related SAEs | 4 | 4 | 1 | 1

3. Primary Outcome: Number of Participants With Grade 3-4 Hematology Abnormalities
Description: Abnormalities were graded per the National Cancer Institute(NCI)Common Toxicity Criteria (CTC), v3.0(Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are as follows: Hemoglobin: Grade 3:6.5 - <8.0g/dL, Grade 4: <6.5g/dL. Platelets: Grade 3: 25.0 - <50.0*10^9/L, Grade 4: <25.0*10. Absolute Neutrophil Count (ANC): Grade 3: 0.5 - <1.0*10^9/L, Grade 4: <0.5*10^9/L.White Blood Cells (WBC) : Grade 3: 1.0 - <2.0*10^9/L, Grade 4: <1.0*10^9/L.
Time Frame: as for outcome 1
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15 | 5 | 4
participants
  WBC | 2 | 1 | 0 | 0
  ANC | 3 | 1 | 0 | 2
  Platelet Count | 3 | 1 | 0 | 1
  Hemoglobin | 0 | 1 | 1 | 1

4. Secondary Outcome: Number of Participants With Complete Hematologic Response (CHR)
Description: CHR should meet all of the following criteria: WBC <= Institutional ULN; ANC >= 1000/mm^3 ; Platelets < 450 000/mm^3 , no blasts or promyelocytes in peripheral blood; < 5% myelocytes plus metamyelocytes in peripheral blood; basophils in peripheral blood < 20% and no extramedullary involvement (including no hepatomegaly or splenomegaly). CHR can begin only 14 days after the start of treatment.
Time Frame: Pre-treatment to study discontinuation. Median duration of exposure (on-study time) was 23.4 months.
Population: All treated participants. Data was not analyzed and reported for the other two groups (Accelerated Phase CML and Myeloid Blast Phase CML) due to small sample sizes.
Measure: Number; unit: participants
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15 | 0 | 0
participants | 16 [49.8 to 89.3] | 13 [59.5 to 98.3] |  |

5. Secondary Outcome: Median Number of Months of CHR (Kaplan Meier Method)
Description: CHR: WBC<=ULN (range: 9.29-12.5*10^3 c\uL); ANC >=1000/mm^3;Platelets <450000/mm^3,no blasts/promyelocytes in peripheral blood; <5% myelocytes+metamyelocytes in peripheral blood; basophils in peripheral blood <20% & no extramedullary involvement. Duration computed for chronic phase participants, measured in months from first day CHR criteria met, provided they are confirmed 4 weeks later, until progression of disease, treatment discontinuation due to progressive disease or death. Participants who neither discontinue due to progression, nor progress nor die censored on date of last assessment.
Time Frame: Pre-treatment to study discontinuation. Median duration of exposure (on-study time) was 23.4 months.
Population: All treated participants with CML (whether QD or BID dosing), who had CHR. Data were not analyzed and reported for the other two groups (Accelerated Phase CML and Myeloid Blast Phase CML) due to small sample sizes.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Participants With Chronic Myelogenous Leukemia (CML): Participants continued on the last dose and schedule of dasatinib that was received within the previous protocol CA180002 (NCT00064233). QD dosing: TDD of 50 mg, 75 mg, 105 mg, 140 mg or 180 mg dasatinib was taken QD. BID dosing: Treatment was received BID, with a TDD of 50 mg, 70 mg, 100 mg, 140 mg, 180 mg or 240 mg dasatinib. Participants were dosed on 1 of 3 schedules: 5 days on, 2 days off; 6 days on, 1 day off; or continuous daily dosing and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
Arm/Group | Participants With Chronic Myelogenous Leukemia (CML)
Number analyzed (Participants) | 29
months | 52.0 [31.9 to NA] — Not reached. Upper limit of the confidence interval was not estimable because not enough subjects had progression subsequent to achieving response.

6. Secondary Outcome: Number of Participants With Major Cytogenetic Response (MCyR)
Description: Cytogenetic responses are based on the prevalence of Philadelphia chromosome positive (Ph+) metaphases among cells in metaphase on a bone marrow sample. MCyR is defined as number of participants with Complete Cytogenetic Response (CCyR): 0% Ph+ cells in metaphase in bone marrow or Partial Cytogenetic Response (PCyR): >0% to 35% Ph+ cells in metaphase in bone marrow.
Time Frame: Pre-treatment to study discontinuation. Median duration of exposure (on-study time) was 23.4 months.
Population: All treated participants with evaluable sample sizes. Data was not analyzed and reported for the Accelerated Phase CML and Myeloid Blast Phase CML groups due to small sample sizes, which would lead to response rate estimates that are not stable.
Measure: Number; unit: participants
Groups:
- Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry: Participants continued on the last dose and schedule of dasatinib that was received within the previous protocol CA180002 (NCT00064233). A total daily dose (TDD) of 50 mg, 75 mg, 105 mg, 140 mg or 180 mg dasatinib was taken once daily (QD). Participants were dosed on 1 of 3 schedules (5 days on, 2 days off; 6 days on, 1 day off or continuous daily dosing) and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
- Participants With CML: BID Dosing at Study Entry: Participants continued on the last dose and schedule of dasatinib that was received within the previous protocol CA180002 (NCT00064233). Treatment was received BID, with a TDD of 50 mg, 70 mg, 100 mg, 140 mg, 180 mg or 240 mg dasatinib. Participants were dosed on 1 of 3 schedules (5 days on, 2 days off; 6 days on, 1 day off or continuous daily dosing) and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | Participants With CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15
participants | 13 | 9

7. Primary Outcome: Number of Participants With Grade 3-4 Serum Chemistry Abnormalities
Description: Abnormalities were graded per the NCI (CTC), v3.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are as follows: Alanine aminotransferase (ALT): Grade 3: 5.0-20.0 * ULN (upper limit of normal), Grade 4: >20.0 * ULN; Calcium: Grade 3: 6.0-<7.0 or >12.5-13.5 mg/dL, Grade 4: <0.6->13.5 mg/dL; Bilirubin: Grade 3: >3-10 * ULN, Grade 4: >10 * ULN; Creatinine: Grade 3: >3.0-6.0 * ULN, Grade 4: >6.0 * ULN; Albumin: Grade 3: <2g/dL (Grade 4 not defined in NCI CTC); Magnesium: Grade 3: 0.6-<0.8 or >2.46-6.6mEq/L, Grade 4: <0.6 or >6.6mEq/L.
Time Frame: as for outcome 1
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15 | 5 | 4
participants
  Low Albumin | 1 | 0 | 0 | 0
  High ALT | 1 | 1 | 0 | 0
  High Total Bilirubin | 0 | 0 | 0 | 0
  Low Calcium | 0 | 0 | 0 | 0
  Low Magnesium | 0 | 0 | 0 | 0
  High Serum Creatinine | 0 | 0 | 0 | 0

8. Secondary Outcome: Median Number of Months of Major Cytogenetic Response (MCyR)
Description: MCyR: 0% Ph+ cells in metaphase in bone marrow or Partial Cytogenetic Response (PCyR): >0% to 35% Ph+ cells in metaphase in bone marrow.The duration of MCyR was computed for chronic phase participants whose best response is either CCyR or PCyR. It was measured in months from the time measurement criteria are first met for CCyR or PCyR (whichever status is recorded first) until the date of progression or death. Participants who neither progress nor die are censored on the date of their last cytogenetic assessment.
Time Frame: Pre-treatment to study discontinuation. Median duration of exposure (on-study time) was 23.4 months.
Population: All treated participants with CML (whether QD or BID dosing), who had MCyR (13 participants had MCyR in QD group and 9 in BID group). Data were not analyzed and reported for the other two groups (Accelerated Phase CML and Myeloid Blast Phase CML) due to small sample sizes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Chronic Myelogenous Leukemia (CML)
Number analyzed (Participants) | 22
months | 50.1 [27.1 to 50.1]

9. Primary Outcome: Number of Participants With Dose Interruptions and Dose Reductions
Description: Dose interruptions and reductions were allowed, in order to optimize individual participant's hematologic, cytogenetic, and molecular response while maintaining and evaluating safety and tolerability of long-term exposure to dasatinib. A dose reduction is defined as the administration of a dose at a lower level compared to previous dose and such that reduced dose, or a lower dose, is given at least 4 consecutive times. In determining the reductions, dose level would be compared to the previous non-null dose. Dose interruption is defined as a complete omission of dosing for 4 consecutive times.
Time Frame: From start of study to final assessment (up to 32.2 months).
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | CML: BID Dosing at Study Entry | Accelerated Phase CML: BID Dosing at Study Entry | Myeloid Blast Phase CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15 | 5 | 4
participants
  Dose interruptions | 7 | 9 | 2 | 2
  Dose reductions | 8 | 4 | 2 | 1

10. Secondary Outcome: Number of Participants With Best Cytogenetic Response
Description: Cytogenetic responses are based on the prevalence of Ph+ metaphases among cells in metaphase on a bone marrow sample. CCyR: 0% Ph+ cells in metaphase in bone marrow, PCyR: >0% to 35% Ph+ cells in metaphase in bone marrow, Minor CyR: >35% to 65% Ph+ cells in metaphase in bone marrow, Minimal CyR: >65% to 95% Ph+ cells in metaphase in bone marrow and No CyR: >95% to 100% Ph+ cells in metaphase in bone marrow.
Time Frame: Pre-treatment to study discontinuation. Median duration of exposure (on-study time) was 23.4 months.
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Chronic Myelogenous Leukemia (CML): QD Dosing at Study Entry | Participants With CML: BID Dosing at Study Entry
Number analyzed (Participants) | 22 | 15
participants
  Complete (0%) | 10 | 7
  Partial (1-35%) | 3 | 2
  Minor (36-65%) | 0 | 1
  Minimal (66-95%) | 3 | 1
  No response | 4 | 3
  Unable to determine | 2 | 1

11. Secondary Outcome: Median Number of Months of Progression-free Survival (PFS) (Kaplan Meier Method)
Description: Interval between randomization date & earliest date of disease progression/death due to any cause, assessed by the Independent Radiology Review Committee (IRRC) using modified World Health Organization (WHO) criteria to define progressive disease (PD): >=25% increase in sum of products of diameters (SOPD) of lesions compared with smallest SOPD recorded for study period or progression of any non-index lesion/appearance of new lesion. If no progression/death, date of last tumor assessment used. For participants who had no on-study tumor assessments & were still alive, date of randomization used.
Time Frame: Baseline to study discontinuation. Median duration of exposure (on-study time) was 23.4 months.
Population: All treated participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Participants: All participants treated in each arm of the study were included.
Arm/Group | All Participants
Number analyzed (Participants) | 46
months | 32.0 [29.8 to NA] — Not reached. Upper limit of the confidence interval was not estimable because not enough subjects had progression event at the time of analysis.

12. Secondary Outcome: Median Number of Months of Overall Survival (OS) (Kaplan Meier Method)
Description: Overall survival was defined as the median number of months from baseline to death from any cause.
Time Frame: Baseline to study discontinuation. Median duration of exposure (on-study time) was 23.4 months.
Population: All treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 46
months | NA [52.8 to NA] — Median and upper limit of confidence interval were not estimable because not enough participants had died at the time of analysis.

ADVERSE EVENTS:
Description: The SAEs listed here differ from those present in the Outcome Measures. This is because the Outcome Measures present on-treatment SAEs and this section presents all SAEs. In addition, the AEs presented here differ from those in the Outcome Measures. This is because the AEs presented here do not include SAEs.
Groups:
- Participants With Accelerated Phase CML; Participants With Myeloid Blast Phase CML: Participants continued on the last dose and schedule of dasatinib that was received within the previous protocol (CA180002; NCT00064233). A TDD of 50 mg, 75 mg, 105 mg, 120 mg, 140 mg or 180 mg dasatinib was taken QD or split into 2 doses and taken BID (TDD of 50 mg, 70 mg, 100 mg, 140 mg, 180 mg or 240 mg ). Participants were dosed on 1 of 3 schedules: 5 days on, 2 days off; 6 days on, 1 day off; or continuous daily dosing and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
- Participants With Chronic Myelogenous Leukemia(CML);QD Dosing: Participants continued on the last dose and schedule of dasatinib that was received within the previous protocol (CA180002; NCT00064233). A total daily dose (TDD) of 50 mg, 75 mg, 105 mg, 140 mg or 180 mg dasatinib was taken once daily (QD). Participants were dosed on 1 of 3 schedules: 5 days, on 2 days off; 6 days on, 1 day off; or continuous daily dosing. Participants were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to twice daily (BID) dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
- Participants With CML; BID Dosing: Participants continued on the last dose and schedule of dasatinib that was received within the previous protocol (CA180002; NCT00064233). Treatment was received BID, with a TDD of 50 mg, 70 mg, 100 mg, 140 mg, 180 mg or 240 mg. Participants were dosed on 1 of 3 schedules: 5 days on, 2 days off; 6 days on, 1 day off; or continuous daily dosing and were permitted to escalate or reduce by 1 dose level at a time, switch from QD dosing to BID dosing and vice versa provided they did not exceed a change of 1 dose level from the TDD. The weekly schedule was also permitted to be increased or decreased 1 level at a time.
Arm/Group | Participants With Accelerated Phase CML | Participants With Chronic Myelogenous Leukemia(CML);QD Dosing | Participants With CML; BID Dosing | Participants With Myeloid Blast Phase CML
Serious Adverse Events (participants affected / at risk) | 3/5 | 10/22 | 9/15 | 3/4
Other Adverse Events (participants affected / at risk) | 5/5 | 21/22 | 15/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Accelerated Phase CML (N=5) | Participants With Chronic Myelogenous Leukemia(CML);QD Dosing (N=22) | Participants With CML; BID Dosing (N=15) | Participants With Myeloid Blast Phase CML (N=4)
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 0 | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 3 | 2 | 1
UROSEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
MENINGITIS (Infections and infestations) | 0 | 1 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 0
CATHETER SITE CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
HERPES ZOSTER DISSEMINATED (Infections and infestations) | 0 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TRANSFUSION-RELATED ACUTE LUNG INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
DEATH (General disorders) | 0 | 2 | 1 | 0
HERNIA (General disorders) | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 1 | 0 | 0
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BLAST CELL PROLIFERATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Accelerated Phase CML (N=5) | Participants With Chronic Myelogenous Leukemia(CML);QD Dosing (N=22) | Participants With CML; BID Dosing (N=15) | Participants With Myeloid Blast Phase CML (N=4)
EYE PRURITUS (Eye disorders) | 0 | 0 | 1 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 1 | 0
OCULAR HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 1
CARDIAC MURMUR (Investigations) | 0 | 2 | 2 | 0
BLOOD CREATININE (Investigations) | 0 | 0 | 1 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 1 | 0
CHEST X-RAY ABNORMAL (Investigations) | 0 | 2 | 0 | 0
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 3 | 1 | 0
ALANINE AMINOTRANSFERASE (Investigations) | 0 | 0 | 1 | 0
BLOOD CHLORIDE INCREASED (Investigations) | 0 | 0 | 1 | 0
BLOOD URIC ACID INCREASED (Investigations) | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 1 | 0
CARDIAC DISORDER (Cardiac disorders) | 0 | 0 | 0 | 1
DILATATION ATRIAL (Cardiac disorders) | 1 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 1 | 0
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 1 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0 | 0 | 0
PALLOR (Vascular disorders) | 1 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0
VASCULAR CALCIFICATION (Vascular disorders) | 0 | 0 | 1 | 0
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 4 | 0
DIZZINESS (Nervous system disorders) | 0 | 2 | 2 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 4 | 0
VOMITING (Gastrointestinal disorders) | 0 | 4 | 3 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 4 | 3 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 1 | 0
GINGIVITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 2 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 1 | 0
DIVERTICULUM (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 1 | 0
SWOLLEN TONGUE (Gastrointestinal disorders) | 0 | 1 | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 1
STOMACH DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 1 | 0
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 3 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 1 | 0
MASTITIS (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 6 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 2 | 1 | 1
BRONCHITIS (Infections and infestations) | 0 | 2 | 2 | 0
HEPATITIS B (Infections and infestations) | 0 | 2 | 1 | 0
ORAL HERPES (Infections and infestations) | 0 | 2 | 0 | 0
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 1
LYME DISEASE (Infections and infestations) | 0 | 2 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 2 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 1 | 1
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1 | 0 | 0 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 2 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 1 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 3 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 5 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
MASS (General disorders) | 0 | 0 | 1 | 0
POLYP (General disorders) | 0 | 0 | 1 | 0
CHILLS (General disorders) | 0 | 2 | 0 | 0
FATIGUE (General disorders) | 1 | 10 | 3 | 2
PYREXIA (General disorders) | 1 | 3 | 2 | 1
ASTHENIA (General disorders) | 0 | 2 | 1 | 0
CALCINOSIS (General disorders) | 0 | 0 | 1 | 0
CHEST PAIN (General disorders) | 1 | 1 | 0 | 0
CHEST DISCOMFORT (General disorders) | 0 | 2 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 4 | 1 | 2
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.